CLINICAL TRIAL: NCT06344741
Title: Comparison of Maternal and Neonatal Outcomes of Early and Late Admission to the Delivery Room
Brief Title: Consequences of Admission to the Delivery Room in the Early and Late Phases
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Assistant Professor, Kocaeli University
Other Study IDs: sdilek6
Record Dates: First submitted 2024-03-21; First posted 2024-04-03 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-06

CONDITIONS: Fear of Childbirth; Neonatal; Pain; Maternal Distress (During Labor); Satisfaction
Keywords: Childbirth; Maternal; Phases
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Latent phase: Participants admitted to the delivery room in the latent phase will be included.
  Interventions: Behavioral: Accepted in latent phase
- Active phase: Participants accepted to the delivery room in the active phase will be included.
  Interventions: Behavioral: Accepted in active phase

INTERVENTIONS:
Behavioral: Accepted in latent phase — Participants admitted to the delivery room in the latent phase will be included. Routine procedures will be performed.
  Other Names: Latent phase
  Groups: Latent phase
Behavioral: Accepted in active phase — Participants admitted to the delivery room in the active phase will be included. Routine procedures will be performed.
  Other Names: Active phase
  Groups: Active phase

SUMMARY:
This study will be conducted to compare maternal and neonatal outcomes of pregnant women who applied to the delivery room in the early (latent) and late (active) phase. The population of the research will consist of participants who applied to Darıca Farabi Training and Research Hospital for birth. To determine the sample size of the study, first, those who meet the inclusion criteria and are admitted to the delivery room in the latent phase and those who are accepted in the active phase will be numbered and recruited sequentially. When the number of participants in the 100 latent and 100 active acceptance groups is reached, the effect size will be calculated using the STAI score averages and the G*Power program, and the exact sample number will be determined, taking into account possible data losses. If necessary, data collection will continue until the target number is reached. Randomization will not be applied in the study. Data will be collected with the maternal and neonatal information form, State and Trait Anxiety Scale (STAI), Fear of Birth Scale, Neonatal Pain and Stress Assessment Scale (ALPS-Neo) and Visual analog scale for birth satisfaction. Data will be collected by the assistant researcher. Statistical analysis will be performed using IBM SPSS Statistic. Descriptive statistical methods will be used to evaluate socio-demographic data, and parametric/nonparametric tests will be used for comparative analyses.

DETAILED DESCRIPTION:
Aim: This study will be conducted to compare maternal and neonatal outcomes of pregnant women who applied to the delivery room in the latent and active phase.

Research hypothesis:

H1.1: There is a statistical difference between the two groups in terms of maternal outcomes of pregnant women who applied to the delivery room in the latent phase and pregnant women who applied in the active phase.

H1.2: There is a statistical difference between the two groups in terms of neonatal outcomes of pregnant women who applied to the delivery room in the latent phase and pregnant women who applied in the active phase.

H0.1: There is no statistical difference between the two groups in terms of maternal outcomes of pregnant women who applied to the delivery room in the latent phase and pregnant women who applied in the active phase.

H0.2: There is no statistical difference between the two groups in terms of neonatal outcomes of pregnant women who applied to the delivery room in the latent phase and pregnant women who applied in the active phase.

Type of Study: This study is a cross-sectional and analytical study planned to compare maternal and neonatal outcomes of pregnant women admitted to the delivery room in the latent and active phases.

The population of the research will consist of participants who applied to Darıca Farabi Training and Research Hospital for birth. To determine the sample size of the study, first, those who meet the inclusion criteria and are admitted to the delivery room in the latent phase and those who are accepted in the active phase will be numbered and recruited sequentially. When the number of participants in the 100 latent and 100 active acceptance groups is reached, the effect size will be calculated using the STAI score averages and the G*Power program, and the exact sample number will be determined, taking into account possible data losses. If necessary, data collection will continue until the target number is reached. Randomization will not be applied in the study.

Data will be collected with the maternal and neonatal information form, State and Trait Anxiety Scale (STAI), Fear of Birth Scale, Neonatal Pain and Stress Assessment Scale (ALPS-Neo).

Maternal and neonatal information form: It was prepared by the researcher within the framework of the literature. The form consists of 49 questions including maternal and neonatal introductory characteristics.

State and Trait Anxiety Inventory (STAI): This scale, developed by Spielberger et al., consists of two subscales: state and continuous, each consisting of 20 questions. It is a Likert-type scale with points between 1 and 4 for each question and can be applied to individuals over the age of 14.

Neonatal pain and stress rating scale (ALPS-Neo): Lundqvist et al. to evaluate pain and stress in premature and term newborns. The Cronbach's alpha coefficient of the scale was reported as 0.95. The scale is a 0-1-2, 3-point Likert-type scale consisting of 5 items in one dimension, including the newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made by observation. A minimum of 0 and a maximum of 10 points are obtained from the scale. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress. The higher the stress and pain, the higher the score.

Fear of Birth Scale: Scale Wijma et al. It was developed to measure fear during birth. The scale is one-dimensional and consists of a total of 10 items. Responses to each item in the scale range from 1 to 10, with 1 indicating "I completely disagree" and 10 indicating "I completely agree". The minimum score that can be obtained from the scale is 10 and the maximum score is 100. A high score from the scale indicates high fear. Five items in the scale (1, 3, 5, 7, and 10) have a positive meaning, and five items (2, 4, 6, 8, and 9) have a negative meaning.

Visual analog scale for birth satisfaction: It consists of 10 cm analog line. How satisfied were you with your birth? 0 was defined as 'I was not satisfied at all' and 10 was defined as 'I was very satisfied'. The participant is asked to mark the appropriate point. It will be filled after birth.

Statistical analysis will be performed using IBM SPSS Statistic. Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of socio-demographic data. When the data is found to be suitable for normal distribution, it will be analyzed with parametric tests (chi-square, T test, etc.) in comparing categorical variables, and when it is not found to be suitable for normal distribution, it will be analyzed with non-parametric tests (Mann-Whitney U Test, Kruskal Wallis, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over,
* At term gestational age (37-42 weeks),
* Does not have a risky pregnancy,
* Single pregnancy,
* Head presentation,
* Literate participants will be included

Exclusion Criteria:

* Those who do not have sufficient mental health to fill out the survey form,
* Visual, hearing, perception impaired
* The newborn is unhealthy or stillborn,
* With membrane rupture
* Having a history of cesarean section
* Those who have contraindications for vaginal birth
* Having complaints of pregnancy-related bleeding,
* Any risk of birth (placental abruption, uterine rupture, etc.)
* Willing to leave at any point during the research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant participants
Study Population: Participants who applied to the delivery room during the study period and met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Neonatal pain and stress | 15th minute after birth
  ALPS-Neo: It is a 3-point Likert type scale consisting of 5 items: facial expression of the newborn, breathing pattern, tone of extremities, hand and foot activities and activity level. Measurements are made through observation. As stress and pain increase, the score obtained also increases. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and above 5 points indicate the presence of serious pain and stress.
Birth satisfaction | 5th hour postpartum
  Birth satisfaction will be measured with a 10cm line visual analogue scale. The participant will be asked about her satisfaction with the birth and will be asked to mark his or her satisfaction on a visual analogue scale. The lowest score from the scale is 0, the highest score is 10.

SECONDARY OUTCOMES:
Maternal Anxiety | During the first 10 minutes of the participant's admission to the delivery room
  Maternal anxiety will be measured with the State and Trait Anxiety Inventory (STAI) during contraction monitoring. The scale consists of two subscales: state and continuous, each consisting of 20 questions. It is a Likert-type scale with points between 1 and 4 for each question, and can be applied to individuals over the age of 14. The lowest score from each of the scales is 20 points and the highest score is 80 points.
Fear of Birth | During the first 10 minutes of the participant's admission to the delivery room
  It will be measured with the Fear of Birth Scale during contraction follow-up. Responses to each item in the scale range from 1 to 10, with 1 indicating "I completely disagree" and 10 indicating "I completely agree". The minimum score that can be obtained from the scale is 10 and the maximum score is 100. A high score from the scale indicates high fear.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D., Study Director — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Lundqvist P, Kleberg A, Edberg AK, Larsson BA, Hellstrom-Westas L, Norman E. Development and psychometric properties of the Swedish ALPS-Neo pain and stress assessment scale for newborn infants. Acta Paediatr. 2014 Aug;103(8):833-9. doi: 10.1111/apa.12672. Epub 2014 May 26. PMID 24813238